CLINICAL TRIAL: NCT02820883
Title: A Single-center, Dose-escalation, Open-label Pilot Study to Evaluate the Safety and Tolerability of a Recombinant Staphylococcus Aureus Vaccine (Escherichia Coli) in Healthy Adults Aged 18-65 Years in China
Brief Title: A Study of a Recombinant Staphylococcus Aureus Vaccine (Escherichia Coli) in Healthy Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Chengdu Olymvax Biopharmaceuticals Inc. (Industry); Third Military Medical University (Other)
Responsible Party: Principal Investigator, Fengcai Zhu, Professor, Jiangsu Province Centers for Disease Control and Prevention
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT027a
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Staphylococcus Aureus Infection
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dosage vaccine (Experimental): High dosage of Staphylococcus aureus vaccine (60µg/0.6ml)
  Interventions: Biological: Staphylococcus aureus vaccine (60µg/per protein)
- Middle dosage vaccine (Experimental): Middle dosage of Staphylococcus aureus vaccine (30µg/0.6ml)
  Interventions: Biological: Staphylococcus aureus vaccine (30µg/per protein)
- Low dosage vaccine (Experimental): Low dosage of Staphylococcus aureus vaccine (15µg/0.6ml)
  Interventions: Biological: Staphylococcus aureus vaccine (15µg/per protein)

INTERVENTIONS:
Biological: Staphylococcus aureus vaccine (60µg/per protein) — two doses of 60µg/0.6ml per dose
  Arms: High dosage vaccine
Biological: Staphylococcus aureus vaccine (30µg/per protein) — two doses of 30µg/0.6ml per dose
  Arms: Middle dosage vaccine
Biological: Staphylococcus aureus vaccine (15µg/per protein) — two doses of 15µg/0.6ml per dose
  Arms: Low dosage vaccine

SUMMARY:
This is an open-label, dose-escalation pilot study with a total of 30 participants with 10 per dosage group. The aim of the pilot study is to explore the preliminary safety of an experimental recombinant staphylococcus aureus vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 to 65 years (aged over 18 and under 66 years).
* Able to comply with all clinical trial protocol requirements and willing to complete all the visit plan process during the whole clinical trial observation period.
* Able to understand the content of informed consent and willing to sign the informed consent.
* Able to complete the diary card independently.
* For females only (18-49 years), a negative urine pregnancy test and willing to practice continuous effective contraception during the study.
* Axillary temperature ≤37.0°C.

Exclusion Criteria:

First Immunization exclusion standard:

* Prior receipt of Staphylococcus aureus vaccine
* Any confirmed Staphylococcus aureus infection disease in the past 12 month.
* History of asthma, hereditary angioneurotic edema, diabetes, malignancy or other serious disease. Participation in the clinical trial is likely to increase the disease risk and interfere with the observation of clinical trial index.
* Prior blood donation or Blood loss over 400ml in the last 3 months;
* Coagulation disorders (coagulation factor deficiency, coagulopathy or platelet disorder) diagnosed by doctors, or obvious bruises or blood coagulation noticed.
* History of allergic disease likely to be exacerbated by any component of the vaccine, including allergy, urticaria, respiratory difficulty, angioneurotic edema or abdominal pain.
* Any autoimmune disease or immunodeficient state, parents, brother and sister with autoimmune disease or immunodeficient disease.
* Taking immunoglobulins and/or any blood products within the last 12 months.
* Asplenia, functional asplenia or asplenia caused by any situation or splenectomy.
* Any acute disease or acute attack of chronic disease in last 7 days.
* History of thyroidectomy or thyroid disease requiring treatment in the last 12 months.
* Immunosuppressor, cytotoxic therapy, inhaled corticosteroid (excluding corticosteroids spray treatment of allergic rhinitis, acute and non-concurrent corticosteroids treatment)
* Participation in another research study involving receipt of an investigational product in the last 30 days.
* Woman who is breast-feeding.
* Prior administration of attenuated vaccine in last 28 days.
* Prior administration of subunit vaccine, inactivated vaccine or allergic therapy in last 14 days.
* Current anti-tuberculosis prophylaxis or therapy
* Any other conditions may compromise the safety or availability of participants in the judgment of the investigator.

Following Immunization exclusion standard:

* Any grade 3 or more serious adverse reaction happen since the last vaccination.
* Other condition violates the inclusion criteria or meets the exclusion criteria is noticed after the first immunization.
* Acute or chronic infections at the vaccination day (axillary temperature>37.0°C).
* According to the investigator, the participant should not continue participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited adverse reactions after vaccination. | within 0-14 days after the vaccination
  Occurrence of solicited site adverse reactions within 0-14 days after vaccination with the Recombinant Staphylococcus aureus vaccine (Escherichia coli).

SECONDARY OUTCOMES:
Occurrence of unsolicited adverse reactions after vaccination. | within 0-35 days after the vaccination
  Occurrence of unsolicited adverse reactions within 0-35 days after vaccination with the Recombinant Staphylococcus aureus vaccine (Escherichia coli).
Occurrence of serious adverse events after the vaccination. | within 6 months after the vaccination
  Occurrence of serious adverse events within 6 months after the vaccination with the Recombinant Staphylococcus aureus vaccine (Escherichia coli).
Changes of the laboratory examinations after vaccination. | day 3 after the vaccination
  Changes of the laboratory examinations after vaccination with the Recombinant Staphylococcus aureus vaccine (Escherichia coli) on day 3.
Changes of the laboratory examinations after vaccination. | day 7 after the vaccination
  Changes of the laboratory examinations after vaccination with the Recombinant Staphylococcus aureus vaccine (Escherichia coli) on day 7.
Changes of the laboratory examinations after vaccination. | day 10 after the vaccination
  Changes of the laboratory examinations after vaccination with the Recombinant Staphylococcus aureus vaccine (Escherichia coli) on day 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Taixing county disease control and prevention, Taishing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes